CLINICAL TRIAL: NCT00127777
Title: Randomized, Multi-Center, Partially Placebo-Controlled Phase IV-Study to Compare Efficacy and Tolerability of 48-Week Combined Therapy With Peginterferon Alfa-2a, Ribavirin and Amantadine Sulphate Versus Placebo in Untreated Patients With Chronic Hepatitis C Virus-Genotype-1-Infection
Brief Title: Peginterferon Alfa-2a, Ribavirin, Amantadine/Placebo in Hepatitis C Virus (HCV)-Genotype-1-Infection (PRAMA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Saarland (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ML17002
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2005-08-25 (Estimated); Status verified 2005-08

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV genotype 1; peginterferon alfa-2a; ribavirin; amantadine; treatment-naive
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine sulphate (in addition to standard treatment)

SUMMARY:
This was a randomized, multi-center, partially placebo-controlled Phase IV study to compare the efficacy and tolerability of a 48-week combined therapy with pegylated interferon alpha-2a, ribavirin and amantadine sulphate versus placebo in untreated patients with chronic hepatitis C virus-genotype-1-infection. The hypothesis was that there will be an increase in sustained response rate for triple therapy compared to current standard treatment.

DETAILED DESCRIPTION:
Primary Objective:

* Proof that a triple-therapy (peginterferon alfa-2a, ribavirin and amantadine sulphate) dispensed over a period of 50 weeks, improves the permanent virological efficacy by more than 10% as compared to a combination therapy with peginterferon alpha-2a and ribavirin, defined as negative HCV-RNA result obtained by a molecular verification method (e.g. Roche AmplicorTM HCV, v.2.0, sensitivity <50 IE/ml) 24 weeks after the end of the therapy.

Secondary Objectives:

* Verification of the initial virological efficacy up to week 12, defined as negative HCV-RNA test results by means of quantitative proof methods, e.g. Roche AmplicorTM HCV Monitor v.2.0 (sensitivity <600 IE/ml).
* Biochemical efficacy, defined by the serum GPT values 24 weeks after the end of the therapy.
* Virological efficacy, measured on the basis of the HCV-RNA values at the end of the therapy.
* Biochemical efficacy defined by the serum GPT values at the end of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects over 18 years of age and below 70 years of age
* Serological indication of chronic hepatitis C infection with positive anti-HCV test and serum HCV-RNA quantification >600 IE/ml by means of quantitative proof methods, e.g. Roche AmplicorTM HCV Monitor test, v.2.0.
* Untreated patients with HCV-induced chronic infection.
* Indication of a genotype HCV-1 on the basis of the reverse hybridizing assay Inno LiPA from Bayer Versant (Innogenetics).
* Increased GPT serum level on at least one determination date within the 56-day screening phase prior to start of administration of study medication.
* Histological identification of inflammatory activity in the liver, with or without an indication of compensated cirrhosis, during the 24 months prior to start of the study.
* Compensated liver disease (Child-Pugh Grade A).
* Negative urine or serum pregnancy test in fertile female subjects within 24 hours before taking the first dose of study medication.
* During the administration of study medication and for 24 weeks after the treatment has stopped, patients must apply two approved contraception methods, one of which must have a barrier effect on the male, e.g. condom.

If one or more of the above inclusion criteria are not fulfilled, the patient is excluded from the study!

Exclusion Criteria:

* Any known sensitive reaction to interferon, ribavirin or amantadine sulphate.
* Pregnant or breast-feeding women and fertile women who do not practice contraception.
* Male partners of pregnant women.
* Previous treatment with interferon and/or ribavirin.
* Treatment with systemic anti-neoplastic or immunomodulatory medication (supraphysiologic doses of steroids or radiation included) within the last 6 months prior to the study and throughout the whole study.
* Immunosuppressed/immunocompromised patients.
* Participation in a clinical study within the last three months.
* Infection with HCV genotype-2, -3, -4, -5 or -6.
* Positive indication of HBsAg, HIV antibodies in the screening phase.
* Non-hepatitis C virus-induced chronic hepatitis (e.g. hematochromatosis, autoimmune hepatitis, metabolic or alcoholic liver disease).
* Decompensated liver cirrhosis or liver disease; Child-Pugh Grade B or C; or threshold compensated liver disease.
* Signs of a hepatocellular carcinoma within 2 months before the randomization, coupled with existing or developing cirrhosis.
* History of oesophagus varices haemorrhage.
* Hemoglobin <12 g/dl in female subjects and <13 g/dl in male subjects in the screening phase.
* Subjects with a higher risk of anemia (e.g. thalassemia, spherocytosis, history of gastrointestinal bleeding) or subjects for whom anemia could be a highly potential medical risk.
* Neutropenia <1500 /µl or thrombocytopenia <90,000 /µl diagnosed in the screening phase.
* Serum creatinine >1.5 mg/dl in the screening phase.
* History of severe psychiatric diseases, especially severe depression, whereby severe psychiatric disease is defined as any anti-depressive or anti-psychotic therapy of at least 3 months in the history, or any indication of suicidal inclination or hospitalization caused by a psychiatric disease.
* Epilepsy.
* Autoimmune disease (e.g. inflammatory intestinal diseases, idiopathic thrombocytopenic purpura, lupus erythematosus sclerodermia, severe psoriasis, rheumatoid arthritis, etc.).
* History of thyroid disease, poorly controlled by prescribed medications
* Chronic pulmonary disease with functional restriction.
* History of severe cardiac disease, e.g. cardiac insufficiency New York Heart Association (NYHA) class III or IV; myocardial infarction within the last 6 months; ventricular tachyarrhythmia requiring treatment; unstable angina pectoris; cerebrovascular circulation disorders; or other significant cardiovascular diseases.
* Patients with pacemakers.
* Cardiomyopathy and myocarditis
* Atrioventricular (AV)-block Grade II and III.
* Previously known bradycardia rating under 55 strokes/minute
* Known, lengthy QT-interval (QTc as per Bazett > 420 ms) or recognizable U waves or hereditary QT-syndrome in the family history.
* History of a severe ventricular arrythmia including Torsade de pointes.
* Simultaneous therapy with budipine or other QT-extending medication such as:

  * Certain antiarrhythmias of class IA (e.g. quinidine, disopyramide, procainamide) and class III (such as amiodarone, sotalol);
  * Certain antipsychotics (e.g. thioridazine, chlorpromazine, haloperidol, pimozide);
  * Certain tri- and tetracyclic anti-depressive medications (e.g. amitriptyline);
  * Certain antihistaminic medications (e.g. astemizol, terfenadin);
  * Certain macrolide antibiotics (e.g. erythromycin, clarithromycin);
  * Certain gyrase inhibitors (e.g. sparfloxacin);
  * Azole-antimycotics and other medications such as halofantrine, cotrimoxazol, pentamidine, cisapride or bepridil;
  * Simultaneous treatment with Memantine.
* Morbus Parkinson.
* History of major organ transplantations, with the exception of cornea transplantation.
* Cancer or any other disease, which, in the opinion of the investigator, is an exclusion criterion for the study.
* Evidence of severe retinopathy (e.g. cytomegalovirus [CMV] retinitis or macular degeneration).
* Patients with narrow-angle glaucoma.
* Active drug abuse (excessive alcohol consumption included) within the last year prior to study (with the exception of a prescribed substitute).
* Patients with state of agitation or confusion
* Patients with a history of acute brain syndrome or exogenous psychosis
* Patients are already enrolled in the study.
* Prostate hypertrophy
* Simultaneous administering of diuretics of combination type triamterene/hydrochlorothiazide.
* Unwillingness or incapability to give written consent after receiving medical information; doubts about the proper protection of patient data; and general reluctance to take part in the study and to adhere to the study terms.

If one or more of these exclusion criteria is fulfilled, the patient shall be excluded from the study!

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2002-07; Study Completion 2006-12

PRIMARY OUTCOMES:
Proof that peginterferon alfa-2a, ribavirin and amantadine sulphate over a period of 50 weeks improves the permanent virological efficacy by more than 10% compared to peginterferon alfa-2a and ribavirin

SECONDARY OUTCOMES:
Verification of the initial virological efficacy up to week 12, defined as negative HCV-RNA test results by means of quantitative proof methods, e.g. Roche AmplicorTM HCV Monitor v.2.0 (sensitivity <600 IE/ml)
Biochemical efficacy, defined by the serum GPT values 24 weeks after the end of the therapy
Virological efficacy, measured on the basis of the HCV-RNA values at the end of the therapy
Biochemical efficacy defined by the serum GPT values at the end of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zeuzem, MD, Principal Investigator — Saarland University Hospital